CLINICAL TRIAL: NCT00642408
Title: Prevention of Intrauterine Growth Retardation in Hounde District, Burkina Faso
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Nutrition Tiers Monde, Belgique (Unknown); Centre Muraz (Other)
Responsible Party: Prof. Patrick Kolsteren, head of the Nutrition and Child Health Unit, Institute of Tropical Medicine, Belgium
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IUGR
Record Dates: First submitted 2008-03-13; First posted 2008-03-25 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Multiple Micronutrient Deficiencies During Pregnancy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MMN (Experimental): multiple micronutrient supplements (MMN): UNIMMAP: vitamin A 800µg, vitamin E 10 mg, vitamin D 5 µg, vitamin B1 1.4 mg, vitamin B2 1.4 mg, niacin 18 mg, vitamin B6 1.9 mg, vitamin B12 2.6 µg, folic acid 400 µg, vitamin C 70 mg, iron 30 mg, zinc 15 mg, copper 2 mg, selenium 65 µg, and iodine 150 µg
  Interventions: Dietary Supplement: Multiple micronutrient supplements (MMN)
- IFA (Active Comparator): iron and folic acid (IFA)(iron 60 mg and folic acid 400µg).
  Interventions: Dietary Supplement: IFA

INTERVENTIONS:
Dietary Supplement: Multiple micronutrient supplements (MMN) — Iron and folic acid: iron 60 mg and folic acid 400µg
  Arms: MMN
Dietary Supplement: IFA — Iron and folic acid (IFA)(iron 60 mg and folic acid 400µg).
  Arms: IFA

SUMMARY:
Intrauterine Growth Retardation is the most important determinant of mortality and morbidity in the neonatal period. It is also a very important factor in predicting nutritional status, health and development in childhood. It even influences health in adult life, contributing to the vicious cycle of disease and poverty. The high rate IUGR in DCs represents therefore a major public health problem. Maternal malnutrition is usually assumed to be a major determinant of the problem in these countries. An increasing amount of evidence points to the potential role played by micronutrient deficiencies during pregnancy. The adverse effect on birthweight of maternal iron deficiency anaemia, lack of zinc and lack of iodine have been documented. A similar effect is suspected for Vitamin A, Magnesium, Calcium, Copper,Thiamine, Pyridoxine and Folic acid. It seems that not one specific deficiency alone is responsible for this adverse effect, but rather a combination of them. Therefore, it is expected that covering needs of pregnant women by a multivitamin-mineral supplement will have an effect of public health importance on children's health.

This study has the objective of improving children's health by preventing intrauterine growth retardation through the provision of multivitamin-mineral supplements during pregnancy.

This research includes 2 constituents:

1. a pilot phase during which socio-anthropological, nutritional and epidemiological aspects of IUGR will be assessed through qualitative and epidemiological methods.
2. a double-blind, randomised, placebo-controlled trial, including 1215 pregnant women aimed at testing 3 hypotheses: supplementing pregnant women with a multivitamin-minerals mix will improve fetal growth; improved fetal growth will have a positive effect on health and growth during infancy; covering nutritional needs of lactating women with a multivitamin-minerals mix during 3 months after delivery will improve health and growth of infants.

The trial is planned in Hounde District, Burkina Faso, in collaboration with Centre Muraz, which plays a leader role in research and services providing at the district level and in policy recommendations at the national level. This will ensure that the study findings are incorporated into on-going district programmes with possible replication at the national level. The research lasts from June 2003 to October 2006.

DETAILED DESCRIPTION:
Low birthweight (LBW; birthweight<2500g) is an important predictor of mortality and morbidity in the neonatal period of early postnatal growth and growth during childhood. It is also associated with cognitive and behavioural development in the first years of life,health status during childhood, and adult health and human capital. As much as 16 % of all live births worldwide present a LBW, more than 90% being in low-income countries.Rates are particularly high in Asia and sub-Saharan countries. In Burkina Faso, it is estimated that 19 % of all live births in 1999-2005 were LBW.

In developing countries, most cases of LBW are attributed to intrauterine growth retardation (IUGR) rather than to preterm delivery.Factors interacting with fetal development are numerous. Among them maternal malnutrition, particularly micronutrient deficiencies, and malaria during pregnancy are assumed to be major determinants of IUGR. Dietary surveys have consistently shown that multiple micronutrient deficiencies, rather than single deficiencies, are common. It is therefore expected that providing multiple micronutrients (MMN), instead of iron and folic acid (IFA) as currently recommended by WHO, could have an effect of public health importance on fetal growth and its correlates. The UNICEF/WHO/UNU multiple micronutrient supplement for pregnancy and lactating women (UNIMMAP) was designed by experts and was proposed for field testing. A recent systematic review concluded that additional evidence was needed to establish the effects of maternal MMN supplements on infant and maternal health. The study described here is part of a series of efficacy studies on the effect of the UNIMMAP supplements on pregnancy outcomes.

The study takes place in the health district of Houndé (south-west of Burkina Faso) in the surroundings of 2 health centers (12,000 inhabitants) from June 2003 to October 2006. Houndé is situated in a Sudano-Sahelian climate belt. The diet is essentially cereal-based. In 2004 and 2006, food consumption surveys estimated the average caloric intake during pregnancy at 8.6 MJ and 8.1 MJ during the postharvest and pre-harvest season respectively. Malaria transmission is permanent with seasonal variations. In 2002, the HIV prevalence among consulting pregnant women in the district was estimated at 2 %. The incidence of LBW in term infants was around 17% at the District Hospital in 2000-2001.

The recruitment of participants is community-based. During a preliminary census, houses in the study area are mapped and numbered and a unique identification code allocated to every woman of child-bearing age. Twenty-five locally trained home-visitors visit monthly every compound for early detection of pregnancy and referral to the health center for pregnancy test. Once the pregnancy is confirmed and after extensive explanation of the study purposes and procedures in Bwamu, Moré or Dioula, participants are asked to provide signed consent or thumbprints. There are no exclusion criteria other than planning to leave the area within the next 2 years.

This study is a double-blind, randomized controlled trial, with directly observed drug intake. Pregnant women are randomly assigned to receive either IFA (iron 60 mg and folic acid 400µg) or MMN (UNIMMAP: vitamin A 800µg, vitamin E 10 mg, vitamin D 5 µg, vitamin B1 1.4 mg, vitamin B2 1.4 mg, niacin 18 mg, vitamin B6 1.9 mg, vitamin B12 2.6 µg, folic acid 400 µg, vitamin C 70 mg, iron 30 mg, zinc 15 mg, copper 2 mg, selenium 65 µg, and iodine 150 µg) until 3 months after delivery. Intervention and control micronutrient tablets are identical in appearance and manufactured by Scanpharm (Copenhagen, Denmark) in containers with a letter code (A/B) for each intervention group. This code is kept secret from study participants and study personnel until data analysis. Micronutrients are kept in a cool room until allocation. Vitamin C levels, identified as the most labile component in the MMN, are monitored once a year and found remarkably constant through the trial. Participants are also randomly assigned to receive either malaria weekly chemoprophylaxis (chloroquine 300 mg) versus intermittent preventive treatment (sulphadoxine 1500 mg and pyrimethamine 75 mg once in the 2nd and 3rd trimester). The malaria component will be analysed separately.

In case of maternal illness, appropriate treatments are provided according to national guidelines. Severely anemic women (hemoglobin < 70 g/L, without dyspnea) receive ferrous sulphate (200 mg) + folic acid (0.25 mg) twice daily, during 3 months whatever their allocation group. All participants also receive Albendazole 400 mg in the second and third trimester. In case of malaria episode despite the preventative treatment, quinine (300 mg, 3 times a day) is given during 5 days. Vitamin A (200.000 IU) is given to all women after delivery, in conformity with the national recommendations.

ELIGIBILITY:
Inclusion Criteria:

All the women of child-bearing age (15-44 years) living in the study area (4 100) will be visited monthly to assess early pregnancy and will be invited to participate in the trial.

Exclusion Criteria:

Will be excluded from the study women :

* planning to move outside the district within the 2 years following the start of the trial.
* regularly using a contraceptive method.
* already pregnant at the start of the trial.

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1370 (Actual)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Weight, length and Rohrer index at birth, and gestational duration in single pregnancies. | At birth
Mortality, morbidity and growth during the first year of life | Monthly during infancy

SECONDARY OUTCOMES:
LBW; SGA; thoracic circumference; head circumference; mid-upper arm circumference; hemoglobin concentration in mothers and in newborns; soluble sTfR in cord blood as an iron status indicator; preterm birth; stillbirth; perinatal death | Different depending on mother and child

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Roberfroid, MD, Principal Investigator — ITM Antwerp; Nicolas Meda, MD, Principal Investigator — Head of the Epidemiology Unit in Centre Muraz; Patrick Kolsteren, MD, Study Chair — head of the Nutrition and Child Health Unit in the Institute of Tropical Medicine (ITM, Antwerp, Belgium)
Locations (1):
- Centre Muraz, 2054, Avenue Mamadou KONATE, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Derived] Roberfroid D, Huybregts L, Lanou H, Ouedraogo L, Henry MC, Meda N, Kolsteren P; MISAME study group. Impact of prenatal multiple micronutrients on survival and growth during infancy: a randomized controlled trial. Am J Clin Nutr. 2012 Apr;95(4):916-24. doi: 10.3945/ajcn.111.029033. Epub 2012 Feb 29. PMID 22378724
- [Derived] Roberfroid D, Huybregts L, Lanou H, Habicht JP, Henry MC, Meda N, Kolsteren P. Prenatal micronutrient supplements cumulatively increase fetal growth. J Nutr. 2012 Mar;142(3):548-54. doi: 10.3945/jn.111.148015. Epub 2012 Feb 1. PMID 22298571
- [Derived] Roberfroid D, Huybregts L, Habicht JP, Lanou H, Henry MC, Meda N, d'Alessandro U, Kolsteren P; MISAME Study Group. Randomized controlled trial of 2 prenatal iron supplements: is there a dose-response relation with maternal hemoglobin? Am J Clin Nutr. 2011 May;93(5):1012-8. doi: 10.3945/ajcn.110.006239. Epub 2011 Mar 2. PMID 21367950
- [Derived] Roberfroid D, Huybregts L, Lanou H, Henry MC, Meda N, Kolsteren F P; Micronutriments et Sante de la Mere et de l'Enfant Study (MISAME) Group. Effect of maternal multiple micronutrient supplements on cord blood hormones: a randomized controlled trial. Am J Clin Nutr. 2010 Jun;91(6):1649-58. doi: 10.3945/ajcn.2009.28855. Epub 2010 Apr 7. PMID 20375185
- [Derived] Roberfroid D, Huybregts L, Lanou H, Henry MC, Meda N, Menten J, Kolsteren P; MISAME Study Group. Effects of maternal multiple micronutrient supplementation on fetal growth: a double-blind randomized controlled trial in rural Burkina Faso. Am J Clin Nutr. 2008 Nov;88(5):1330-40. doi: 10.3945/ajcn.2008.26296. PMID 18996870
- See also: Institute of Tropical Medicine Prince Leopold, Antwerp, Belgium — http://www.itg.be